CLINICAL TRIAL: NCT05509283
Title: Nudging Flu Vaccination in Patients at Moderately High Risk for Flu and Flu-related Complications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Collaborators: National Bureau of Economic Research, Inc. (Other); Massachusetts Institute of Technology (Other)
Responsible Party: Principal Investigator, Christopher F Chabris, PhD, Professor, Geisinger Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022-0410
Record Dates: First submitted 2022-08-18; First posted 2022-08-22 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Influenza; Vaccination; Health Promotion; Health Behavior; Risk Reduction
Keywords: Flu Vaccine; Choice Architecture; Machine Learning; Perceived Credibility
MeSH Terms: conditions — Influenza, Human; Health Behavior; Risk Reduction Behavior | interventions — Numbers Needed To Treat

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Providers who prescribe vaccination and diagnose conditions will not be randomized to study arms or informed of patient assignment. Although patients will not be explicitly informed which arm they have been randomized to, they will be aware of the messages they receive.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Passive control (No Intervention): Patients in the passive control arm will receive no additional pro-vaccination intervention beyond the health system's normal efforts. Although some patients are currently targeted for flu vaccination encouragement due to a conventional non-ML assessment that they are at high risk for complications, these patients are not told that they are at high risk or that they have been targeted.
- Active control (Experimental): Patients in the active control arm will receive messages reminding them to get a flu shot without being advised of their risk status.
  Interventions: Behavioral: Risk Reduction
- High risk only (Experimental): Patients in this treatment arm will receive messages telling them they have been identified to be at high risk for flu complications, without specifying how or why the health system believes this to be the case.
  Interventions: Behavioral: Risk Reduction
- Risk based on medical records (Experimental): Patients in this treatment arm will receive messages telling them they have been identified to be at high risk for flu complications via review of their medical records.
  Interventions: Behavioral: Risk Reduction
- High risk based on algorithm (Experimental): Patients in this treatment arm will receive messages telling them they have been identified to be at high risk for flu complications via analysis of their medical records by a computer algorithm.
  Interventions: Behavioral: Risk Reduction

INTERVENTIONS:
Behavioral: Risk Reduction — Letter, patient portal, SMS and/or another modality
  Arms: Active control; High risk based on algorithm; High risk only; Risk based on medical records

SUMMARY:
This study will test the relative efficacy of high-risk messages in increasing flu shot rates in patients at moderately high risk for flu and complications (those in the top 11-20% of risk). It will also examine whether informing patients that their high-risk status was determined by analyzing their medical records or by an artificial intelligence (AI) / machine-learning (ML) algorithm analyzing their medical records will affect the likelihood of receiving a flu vaccine.

DETAILED DESCRIPTION:
Almost everyone age 6 months or older can benefit from the vaccine, which can reduce illnesses, missed work, hospitalizations, and death by reducing the likelihood of contracting influenza. Flu shots are particularly important for patients at high risk of experiencing severe outcomes.

In the 2020-21 and 2021-22 flu seasons, the study team sent messages to Geisinger patients in the top 10% of risk for flu and complications according to an artificial intelligence algorithm. Messages that disclosed patients' risk status significantly increased flu vaccination rates. Additionally, messages that included risk information were most effective in patients at relatively lower risk (those in the top 4-10%) compared with those at the highest risk (top 3%).

The present work will test the effectiveness of high-risk messages in patients who are in the top 11-20% of risk, at high risk but lower than previous studies. These communications will inform patients they are at high risk with either (a) no additional explanation, (b) an explanation that this determination comes from an analysis of their medical records, or (c) the additional explanation that an AI or ML algorithm made this determination.

ELIGIBILITY:
Inclusion Criteria:

* Included on a list of active Geisinger patients (all patients on this list attended at least one primary care appointment at Geisinger between 10/1/2008 and 4/13/2022, and either had a Geisinger primary care provider assigned as of April 2022, or were in the Electronic Health Record [EHR] since at least September 2021 and had at least one encounter in 2020-2022)
* Aged 18 or older
* In the top 11-20% of risk for flu and flu complications, according to Medial's flu complications machine learning algorithm (which operates on coded EHR data)
* Has a Geisinger PCP assigned as of August 2022
* Has had an encounter in the last 2 years as of August 2022

Exclusion criteria:

- Cannot be contacted via any of the communication modalities (e.g., letter, patient portal, SMS) being used in the study, either due to insufficient/missing contact information in the EHR or because they opted out of all modalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40671 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
Flu vaccination | Within 6 weeks of the patient's study start date
  Received a flu vaccination within within 6 weeks of the patient's study start date

OTHER OUTCOMES:
High confidence flu diagnosis | Up to 8 months
  Patient received a flu diagnosis via a positive polymerase chain reaction (PCR)/antigen/molecular test (yes/no) during the 2022-23 flu season (from the patient's study start date through April 30, 2023).
"Likely flu" diagnosis | Up to 8 months
  Received a "high confidence flu" diagnosis (with positive PCR/antigen/molecular test) and/or "likely flu" diagnosis (as assessed via International Classification of Disease [ICD] codes or Tamiflu administration or positive PCR/antigen/molecular test) (yes/no) during the 2022-23 flu season (from the patient's study start date through April 30, 2023).
  Note that "likely flu" is a superset of the "high confidence flu" diagnoses.
Flu complications | Up to 11 months
  Diagnosed with flu-related complications (yes/no) from the patient's study start date through July 31, 2023.
ER visits | Up to 11 months
  Number of ER visits from the patient's study start date through July 31, 2023.
Hospitalizations | Up to 11 months
  Number of hospitalizations from the patient's study start date through July 31, 2023.
COVID-19 vaccination rates | Up to 8 months
  Received at least one COVID-19 vaccination (yes/no) during the 2022-23 flu season (from the patient's study start date through April 30, 2023).

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Chabris, PhD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data with no personally identifiable information will be made available to other researchers on the Open Science Framework for transparency. This will include the essential data and code needed to replicate the analysis that yielded reported findings.
Supporting Information: Study Protocol
Time Frame: The data will become available after publication of study results in a scientific journal and will be available as long as the Open Science Framework hosts the data.
Access Criteria: The data on the Open Science Framework will be open to anyone requesting that information.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-25): https://cdn.clinicaltrials.gov/large-docs/83/NCT05509283/Prot_SAP_000.pdf